CLINICAL TRIAL: NCT04526860
Title: Maternal Obesity Programs Offspring Hypothalamic Neurogenesis and Appetite: Mechanisms and Prevention of Hyperphagia-mediated Childhood Obesity
Brief Title: Determine if Human Infant Weight Gain Can be Modulated to Prevent Obesity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding period ended, impact of Covid
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Michael Ross, Distinguished Professor of Obstetrics & Gynecology, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 31686-01R
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Obesity, Infant
Keywords: obesity, hyperphagia, breast milk
MeSH Terms: conditions — Pediatric Obesity; Obesity; Hyperphagia

STUDY DESIGN:
Intervention Model Description: Calibration of infant breast milk and formula intake: We will calibrate (reduce) the pumped breast milk or formula intake of infants of overweight and obese mothers who exceed 2 standard deviations of normal WHO weight standards, in order to prevent infant obesity and subsequent childhood obesity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Infant Feed Group (No Intervention): Infants will receive human milk or formula milk ad libitum.
- Calibrated Infant Feed Group (Other): Infants will have reduced human milk or formula milk intake.
  Interventions: Other: Calibration of infant breast milk and formula milk intake

INTERVENTIONS:
Other: Calibration of infant breast milk and formula milk intake — We will calibrate (reduce) the pumped breast milk or formula intake of infants of overweight and obese mothers who exceed 2 standard deviations of normal WHO weight standards, in order to prevent infant obesity and subsequent childhood obesity.
  Arms: Calibrated Infant Feed Group

SUMMARY:
The global obesity epidemic has extended to low and middle income countries (LMICs) in which in a dramatic nutritional transition has shifted from maternal/child undernutrition to overnutrition. Within Brazil, maternal overweight/obesity (OW/OB) and childhood obesity have dramatically increased. During developmental periods, exposure to maternal OB and high-fat diet increases the risk of childhood and adult obesity, in part a result of increased food intake. Studies confirm that offspring of overweight and obese (OW/OB) women are at increased risk of newborn and age 1 year adiposity, and infant adiposity predicts childhood and adult obesity. The investigators hypothesize that that infants of OW/OB mothers have both relative increased appetite and are provided human milk with increased caloric composition. The investigators propose that calibrating milk or formula intake in infants of overweight mothers can reduce the incidence of infant obesity.

DETAILED DESCRIPTION:
This is a clinical intervention study to calibrate infant milk or formula intake and modulate infant weight gain to prevent the development of infant obesity. The studies will be performed at the Ana Abrão Breastfeeding Center, Federal University of São Paulo, Brazil.

Postpartum women will be with pre-pregnant BMI 30 who are providing exclusive human milk via pumping and bottle (n = 50; 50 percent male and 50 percent female) will be recruited at the 7-9 week postpartum visit, Study women will be randomly assigned (computer generated; blocks of 10) to a Standard Feed (SF) or Calibrated Feed (CF) groups. Both groups will be seen at 2 week intervals for assessment of infant weight, supine length, BMI and skinfold thickness. Continuation of exclusive human milk will be confirmed with questionnaires.

In the SF group, mothers will provide bottled human milk ad libitum. In the CF group, infant weight will be assessed in relation to the daily milk volume and approximate caloric intake (based upon maternal human milk sample analysis). Should infants be within 10th to 90th percentile of WHO BMI growth curves, no intervention will be made. Should the infant be greater than 90th percentile of WHO BMI, the provided human milk volume and daily calorie intake will be adjusted in relation to previously established normal volumes for newborn age, with the input of pediatric physician. In no case, will the daily milk volume or calorie intake be reduced by more than 10%. At the subsequent visit, adjustments in milk volume and calorie intake will continue, dependent upon the infant BMI trend, accommodating the normal increase in milk intake with advancing age. Should the infant be less than 10th percentile of WHO BMI, the maternal- infant dyad will be referred for a pediatric and nutrition consults to assess the cause and treatment for potential nutrient deficiency. At 26 wks, the investigators will assess the distribution of infant weight BMI between SF and CF groups.

An identical Study will be undertaken (Standard Feed and Calibrated Feed), with the exception that only current formula feed mothers will be enrolled. All women will be provided a standard brand of commercial formula feed, for which total caloric content and composition will be determined.

Data Analysis. The investigators will compare standard feed vs calibrated feed infant BMI curves with repeated measures ANOVA (time, BMI) with covariates of the group assignment. The investigators will compare infant weight and BMI curves by maternal BMI and infant birth weight, and between human milk and formula groups. The investigators will analyze growth curves of infants exceeding WHO standards which received adjustments in feedings to assess if early changes in growth curves or milk composition is predictive of weight changes, so as to determine the potential for interventions prior to 90th percentile.

ELIGIBILITY:
Mother infant dyads are eligible for the study, with equal proportion of male and female infant in each study group.

Inclusion Criteria:

* Breast Milk Calibration Study: Study women (pre-pregnant BMI>30) who are providing exclusive human milk via pumping and bottle (50%/50% male/female) will be recruited at the 7-9 week postpartum visit.
* Formula Milk Calibration Study: Study women (pre-pregnant BMI>30) who are providing formula via bottle (50%/50% male/female) will be recruited at the 7-9 week postpartum visit.

Exclusion Criteria:

* Breast Milk Calibration Study: breast implants, prior breast surgery, flat/ inverted nipples, tongue-tie or low birth weight infants.
* Formula Milk Calibration Study: low birth weight infants.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2026-12-20 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Infant normalized weight at 6 months of age | 6 months
  We will quantify effects of calibrated human milk or formula intake on the normalized weight of infants at 6 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Ross, MD, Principal Investigator — The Lundquist Institute; Mina Desai, PhD, Principal Investigator — The Lundquist Institute
Locations (1):
- Breastfeeding Center Ana Abrao, Federal of São Paulo University, Brazil, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared at national and international meetings spanning obstetrics, pediatrics and public health. The findings of the study will be published according to NIH guideline for publication and accepted manuscripts will be deposited to Pub Med Central to ensure public access.
  For the Brazilian community, we will disseminate research data through educational program, workshops and conferences organized by the Brazil Ministry of Health. It is important to note that we plan to translate our research findings first into Portuguese (language of Brazil) as well as Spanish which is the predominant language spoken in our neighboring countries surrounding Brazil.
Supporting Information: CSR
Time Frame: Data available at completion of protocol estimated Dec 2023
Access Criteria: Established research organization

REFERENCES:
- [Background] Conde WL, Monteiro CA. Nutrition transition and double burden of undernutrition and excess of weight in Brazil. Am J Clin Nutr. 2014 Dec;100(6):1617S-22S. doi: 10.3945/ajcn.114.084764. Epub 2014 Oct 29. PMID 25411303
- [Background] Satpathy HK, Fleming A, Frey D, Barsoom M, Satpathy C, Khandalavala J. Maternal obesity and pregnancy. Postgrad Med. 2008 Sep 15;120(3):E01-9. doi: 10.3810/pgm.2008.09.1920. PMID 18824817
- [Background] Kaul P, Bowker SL, Savu A, Yeung RO, Donovan LE, Ryan EA. Association between maternal diabetes, being large for gestational age and breast-feeding on being overweight or obese in childhood. Diabetologia. 2019 Feb;62(2):249-258. doi: 10.1007/s00125-018-4758-0. Epub 2018 Nov 13. PMID 30421138
- [Background] Davenport MH, Cabrero MR. Maternal nutritional history predicts obesity in adult offspring independent of postnatal diet. J Physiol. 2009 Jul 15;587(Pt 14):3423-4. doi: 10.1113/jphysiol.2009.174896. No abstract available. PMID 19602635
- [Background] Guo SS, Wu W, Chumlea WC, Roche AF. Predicting overweight and obesity in adulthood from body mass index values in childhood and adolescence. Am J Clin Nutr. 2002 Sep;76(3):653-8. doi: 10.1093/ajcn/76.3.653. PMID 12198014
- [Background] Catalano PM. Obesity and pregnancy--the propagation of a viscous cycle? J Clin Endocrinol Metab. 2003 Aug;88(8):3505-6. doi: 10.1210/jc.2003-031046. No abstract available. PMID 12915626
- [Background] Prentice P, Ong KK, Schoemaker MH, van Tol EA, Vervoort J, Hughes IA, Acerini CL, Dunger DB. Breast milk nutrient content and infancy growth. Acta Paediatr. 2016 Jun;105(6):641-7. doi: 10.1111/apa.13362. Epub 2016 Apr 6. PMID 26865238
- [Background] Isganaitis E, Venditti S, Matthews TJ, Lerin C, Demerath EW, Fields DA. Maternal obesity and the human milk metabolome: associations with infant body composition and postnatal weight gain. Am J Clin Nutr. 2019 Jul 1;110(1):111-120. doi: 10.1093/ajcn/nqy334. PMID 30968129
- [Background] Young BE, Levek C, Reynolds RM, Rudolph MC, MacLean P, Hernandez TL, Friedman JE, Krebs NF. Bioactive components in human milk are differentially associated with rates of lean and fat mass deposition in infants of mothers with normal vs. elevated BMI. Pediatr Obes. 2018 Oct;13(10):598-606. doi: 10.1111/ijpo.12394. Epub 2018 Aug 9. PMID 30092608
- [Background] Brunner S, Schmid D, Zang K, Much D, Knoeferl B, Kratzsch J, Amann-Gassner U, Bader BL, Hauner H. Breast milk leptin and adiponectin in relation to infant body composition up to 2 years. Pediatr Obes. 2015 Feb;10(1):67-73. doi: 10.1111/j.2047-6310.2014.222.x. Epub 2014 Apr 14. PMID 24729519